CLINICAL TRIAL: NCT04536909
Title: Indication and Treatment of Adult Kyphoscoliosis
Acronym: INTRAKS
Status: Active, not recruiting | Type: Observational
Sponsor: University of Bergen (Other)
Collaborators: Oslo University Hospital (Other); Kyoto University Hospital (Other); Region Örebro County (Other); Skane University Hospital (Other); Haukeland University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 1126
Record Dates: First submitted 2020-04-27; First posted 2020-09-03 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Kyphoscoliosis
Keywords: deformity; spine; kyphosis; scoliosis
MeSH Terms: conditions — Congenital Abnormalities; Kyphosis; Scoliosis | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-surgical: A non-surgical group for comparison, they will conduct a training program tailored for the kyphoscoliotic patients. The inclusion criteria is the same as for the surgical group.
  Interventions: Other: Non-surgical
- Surgical: Patients operated with correction of kyphotic- or scoliotic deformity.
  Interventions: Procedure: Surgical

INTERVENTIONS:
Other: Non-surgical — We have constructed a training program with help from physiotherapists from Rikshospitalet in Oslo, tailored for kyphotic- and scoliotic patients.
  Groups: Non-surgical
Procedure: Surgical — Surgery for correction of kyphotic- or scoliotic deformity.
  Groups: Surgical

SUMMARY:
Degeneration, iatrogenic-/idiopathic causes and fractures can lead to kypho- scoliotic deformities potentially resulting in pain and loss of function. The surgical strategies rely on surgeon preferences and type of deformity as well as clinical symptoms. The complication rate of surgical treatment is high. The aim of this study is to elucidate the indications for surgical treatment of kyphoscoliosis and evaluate the effectiveness of surgical and non-surgical outcome clinically and radiologically.

The primary outcome for the PROMs and x-ray is at 12 months, but the investigators will also follow the patients with the PROMs and x-rays after 2,5 and 10 years.

DETAILED DESCRIPTION:
Detailed description 1 Indications and Treatment of Adult Kypho- Scoliosis (INTRAKS Study) 2. Background:New surgical techniques for osteotomies and promising equipment has led to a renaissance with broader indications, evoking the need for well-founded studies and quality registration of the adult kyphoscoliosis treatment to evaluate the risk of major complication, the benefit for the patients and socioeconomic burden. Prior randomized studies have had high crossover rates to surgical treatment, questioning the result of the studies. As a randomized controlled trial (RCT) will be difficult, the investigators plan to propensity match two cohorts and then compare the correctional surgery and non- surgical treatment at a 1 year follow-up.

2.1 Needs description:

1. Identify predictors for unsatisfactory outcome in adult kyphoscoliosis. This study aims to create a predictive model for unsatisfactory outcome after deformity surgery in adult kyphoscoliosis. A prospective multicenter observational effectiveness study is constructed to detect a < 30% improvement from baseline in Oswestry Disability Index (ODI) score at 12 months follow up. The predictive model can be a helpful tool in accessing the complexity of this patients and aid in shard decision making and improved surgical planning. Patients are grouped in: 1) unsatisfactory result (UR) < 30% increase from baseline ODI score, 2) satisfactory result (SR) ≥ 30% increase from baseline ODI score. A predictive model will be calculated for both kyphosis and scoliosis together and separately. The same criteria for inclusion are set in the non-surgical group as well as all the data collected, a predictive model will be created if the difference in outcome is significant. The investigators will also look at the patients with a > 10% worsening from baseline in ODI score at 12 months follow up.
2. A prospective multicenter observational effectiveness study of adult kyphoscoliosis treatment, surgical and non-surgical outcome with a 12 months follow up.

   1. This part of the study will be looking at the effectiveness of surgery vs non-surgical treatment using the PROMS described in the protocol. It is outcome related, the planned follow up time is 12 months, but the investigators have ethical approval (REK) to continue the data recording for 24 months and more for a sufficient follow up time. It exceeds the time limit for the PhD candidates listed, but others will continue the work. It will contain all the patients included.
   2. The subgroups of iatrogenic/degenerative kyphosis and scoliosis will be studied separately as it is known that the mainly scoliotic patients do better than the kyphotic once. Around 30-40 patients will be sufficient in each surgical subgroup, the same in the non-surgical.
3. The kyphotic healed high energy fracture. One of the subgroups to be investigated is the high energy fractures healed in kyphosis. High energy fractures are typical males in the age of 25-50. The fractures healed in kyphosis with a regional kyphotic angle of >20 degrees and a positive sagittal vertical axis of >4 cm can be included (the rest of the inclusion or exclusion criteria listed will be followed as for the whole study). As this is a subgroup, around 30-40 surgical patients will be sufficient. The investigators hope to have the same number in the non-surgical group to compare with. The main outcome parameter is ODI, but the investigators will also look into the results of the EQ-5D, SRS22 and the numeric rating scale (NRS). As this is a fracture resulting in a secondary deformity, the PROMS listed should be addressing the patient problems.
4. XLIF vs anterior-/transforaminal interbody fusion/pedicle subtraction osteotomy/Smith Petersen/Ponte (ALIF/TLIF/PSO/SP/Ponte).

   There is a trend towards using XLIF and OLIF procedures for deformity cases. The investigating party will look into the patients operated using the lateral approaches and compare it towards the dorsal applied interventions (TLIF, PSO, Ponte/SP), if possible also ALIF patients. It should be at least 30-40 patients undergoing the lateral intervention to be able to make a comparison that could be statistical significant.
5. Socioeconomic study; surgery vs non-surgical for adult kyphoscoliosis. The correctional surgery is often of long duration with expensive implants and highly complicated with high risk of complications. It is costly and the investigators intend to evaluate the socioeconomic burden. The duration of surgery, cost of implants and duration of hospital stay will be registered, the readmission due to complications will be registered for the first 12 months. As EQ-5D is used as a PROM in this study, it will be used for the socioeconomic study.
6. Identify differences in indication, examination and treatment between a European and Asian population.

   This is an international multicenter study in cooperation with the Kyoto University Hospital in Japan.

   The investigators have already detected some vital differences in the surgical approach for the patient group and further comparison will be of interest. The patients, indications, examination as well as the non-surgical and surgical treatment will be examined.
7. Changes in urination and sexual function in a surgical and non- surgical cohort.

   Few studies address this issue, for spine patients it is of great importance and highly underreported. There are few suitable PROMS, so the investigators will use a PROM from a prior study. It is slightly different for men and women due to the differences in sex and it has no scoring system. It has not been validated, so the outcome will be slightly unsatisfactory, the positive sides convinced us to take use of the non-validated form. The investigators have had it translated into Japanese and Swedish and are interested in the Japanese contribution in regard of their cultural differences.
8. Quality control of the Norwegian Quality Register for Spinal Surgery. The investigators will be conducting x-ray measurements (sagittal vertical axis and pelvic parameters, lumbar lordosis) and compare it with the values that the surgeons have entered into the Norwegian quality register for spinal surgery. The measurements will be conducted by an independent radiologist at Haukeland or Oslo University Hospital in Norway and by the PhD student in Norway. It will be an inter-and intra-observer study. The values mentioned above have been used for the last year in the register and a quality control would be of interest.
9. Spinal stiffness after spinal fusion using the Lumbar spine disability index (LSDI).

The Lumbar spine disability index (LSDI) is developed by our Japanese colleges at the Kyoto University Hospital and they are motivated to test it on the deformity patient. It is the second (2/2) non validated PROMS in this study and have been translated from Japanese to Norwegian and Swedish. It has been published in peer review papers by our Japanese colleges. Most likely it will be of most interest to our Japanese colleges and they will go forward with the publishing of the result.

4. Project methodology 4.1 Project design, method selection and analyses Patients to be operated for the correction of spinal deformity during the following two-tree years at Oslo University Hospital Ullevål in Norway, Haukeland University Hospital in Bergen Norway, Malmö University Hospital in Sweden, Örebro University Hospital in Sweden and Kyoto University Hospital in Japan. A randomized controlled trial (RCT) will be difficult, so the investigators plan to propensity match the two cohorts and compare correctional surgery and non- surgical treatment at 1 year follow-up. During the 1 year follow-up period the non-surgical patients will attend an intensive and structured physio-logical training program.

The patient inclusion will follow at the polyclinic by the surgeon; the patient will be presented to the "Intraks.org" homepage for the study. An information leaflet will be handed out and the patient will be given time to decide. If the patient is eligible to the study and agrees to join, a study number will be created using google Sheet, then the patient will be introduced to the informed consent form, paper form in Sweden and Japan, in Norway it can be signed using "Nettskjema" an "Bank ID". Nettskjema is an internet form used to create questionnaire, it is secure, but not secure enough for sensitive patient data, so the data from the forms will be imported directly to "service for sensitive data" (TSD). TSD is a service from Oslo University, secure for all sensitive data and in use for several prospective studies. In the homepage, the patients will, in addition to the informed consent, find the patient reported outcome measures (PROMS). The home page can be found using smartphone, tablet or computer and all forms can be filled out using the homepage. 12 months after surgery or inclusion to non-surgical treatment, the patient need to fill out the forms again. For the non-surgical treatment the homepage (Intraks.org) contains specific text, illustrations and videos with training instruction for the non-surgical treatment, developed with dedicated physiotherapists from Oslo University Hospital. The training-program consists of 3 levels of muscle core training and stretching to be exercised 1-3 times a week for 12 months. They will have a training diary to follow up the compliance that will be controlled at the 3 months follow up. The exercises are available at intraks.org as illustration, text and video.

See the protocol for detailed data collection. 4.2 Project management See protocol. 4.3 Plan for implementation

See protocol, in addition:

The "intraks.org" homepage will be updating the public on published articles and other activities.

4.4 Statistical analysis Altogether 75-100 patients are expected eligible for inclusion in the surgical group of WP2 annually. For the non-surgical treatment, approximately the same number will be needed. By using alfa=5% and power=80% to detect 30% ODI improvement from baseline and 30% improvement in proportion of patients that improved and calculating for 10% crossover, 10% mismatch in the propensity score matching and sufficient power for the subgroup analyzes, the study will need a total of 300 patients. Considering drop outs, the study would have enough patients after 2-3 years of inclusion.

Predictive analysis: Frequency analyses for categorical variables will be conducted via Pearson's c2 analysis. All analysis will be conducted using commercially available software (SPSS version 24, IBM Inc.) and the level of significance is set to p<0.05 in a two-sided test. For the predictive model, missing values within the database will be imputed using standard techniques such as mean and median imputation. Once a complete data set is constructed, an ensemble of decision trees will be constructed with a binary target variable that includes patients with: 1) unsatisfactory result (UR) < 30% increase from baseline ODI score (code = 0), 2) satisfactory result (SR) ≥ 30% increase from baseline ODI score (code = 1). The decision-tree algorithm is C5.0 and 5 different bootstrapped models will be built. Internal validation is accomplished via a 70/30 data split for training and testing the model, respectively. Final overall predictions from the models will be combined and chosen by voting with random selection for tied votes. Overall accuracy and the area under the receiver operating characteristic (AUROC) curve will be calculated as well as predictor importance as determined by the model. The model will be built using commercially available software (SPSS Modeler version 24, IBM Inc.). A sensitivity analysis will be performed 1-2 years into the study period, the MCID/"satisfactory result" and power will be adjusted accordingly

ELIGIBILITY:
Inclusion Criteria:

* Out of coronar or sagittal balance: A correction of 20 degrees or more is possible due to the degree of degeneration.
* >25 years
* >30% ODI score

Exclusion Criteria:

* Do not want to participate and not able to answer PROMs
* Acute fractures (not healed fractures)
* Disc prosthesis
* Neuromuscular cause of deformity (the investigators include Parkinson patients)
* Activ infection or malignancy
* Ideopatic scoliosis with typical add on (the investigators include those that have <20 degrees of scoliosis at Risser 5 and/or the scoliosis increase in age due to degeneration). If unknown, the patient will be included as a de novo scoliosis.

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients from the age of 25 and older are included in the study, if they have a deformed spine that fulfil the inclusin criteria and non of the exclusion criteria. The patients are selected from the outpatient clinic in the including university hospitals (Area of Kyoto in Japan, Örebro in Sweden and the vestcoast as well as the souteast area of Norway).
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Oswestry Disability Index (ODI) | 12 months
  One of the principal condition-specific outcome measures for spinal disorders. Scale from 0-100%, high scores equales increasing disability; 0-20% minimal disability, 20-40% moderat disability, 40-60% severe disability, 60-80% crippled, 80-100% bed bound or exaggerating their symptoms.

SECONDARY OUTCOMES:
Euroqol (EQ-5D) | 12 months
  Changes in the HRQL measured with the EQ-5D between baseline and 12 Changes in the HRQL measured with the EQ-5D between baseline and 12 month follow up. The EQ-5D 3L VAS scale is numbered from 0 to 100. 100 means the best health the participant can imagine. 0 means the worst health the participant can imagine. The descriptive systeme element of the EQ-5D Questionnaire produces a 5-digit health state profile that represents the level of reported problems on each of the five dimensions of health, e.g. 11223 (mobility, self care, activity, pain, anxiety). The health state may subsequently be converted into a single summary number (index value) which refelcts how good or bad a health state is according to the preference of a general population of country/region.
Numeric rating scale (NRS) | 12 months
  Patient reported leg and back pain on a numeric rating scale from 0-10=maximum pain
Scoliosis research society (SRS22) | 12 months
  Score for deformity- spine. 22 questions, 5=best, 1=worst. Unanswered questions: reduce questions answered denominator by appropriate number. Delete questions with more than one response. Domain can not be answered if fewer than three questions answered for that domain. Each domain has a total sum score ranging from 5 to 25, except for satisfaction, which ranges from 2 to 10. The sum of the first 4 domains gives a maximum subtotal of 100, and when the satisfaction domain is included, the maximum total is 110.
Lumbar stiffness disability index(LSDI) | 12 months
  Stiffness of the lumbar spine and its influence in daily activity, compare before and after surgery. 10 questions, scoring: A-E, A=no influence, B=mild influence, C=moderat influence, D=need help, E=not able. The answers A and B can be described as patients with light symptomes and a % of the total can be calculated to se how influencial av spinal fixation can be regarding lumbar stiffness.
Urination- and sexual function (USF) | 12 months
  Questionnaire for urination and sexual function women/man. The questionnaire is not validated, it has no scoring system. There are differences between man and women leading to unequal questionnaire. It might give us information using one and one answer: some are yes/no, freetext or 3-7 possible answers.

CONTACTS AND LOCATIONS:
Overall Officials: Stephan M Rohrl, PhD, Study Director — Oslo University Hospital Ullevåll
Locations (5):
- Kyoto University Hospital, Kyoto, Japan
- Norway (2):
  - Haukeland University Hospital, Bergen
  - Ullevål University Hospital, Oslo
- Sweden (2):
  - Malmö University Hospital, Malmo, Skåne County
  - Örebro University Hospital, Örebro

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ailon T, Shaffrey CI, Lenke LG, Harrop JS, Smith JS. Progressive Spinal Kyphosis in the Aging Population. Neurosurgery. 2015 Oct;77 Suppl 4:S164-72. doi: 10.1227/NEU.0000000000000944. PMID 26378354
- [Background] Auerbach JD, Lenke LG, Bridwell KH, Sehn JK, Milby AH, Bumpass D, Crawford CH 3rd, O'Shaughnessy BA, Buchowski JM, Chang MS, Zebala LP, Sides BA. Major complications and comparison between 3-column osteotomy techniques in 105 consecutive spinal deformity procedures. Spine (Phila Pa 1976). 2012 Jun 15;37(14):1198-210. doi: 10.1097/BRS.0b013e31824fffde. PMID 22366971
- [Background] Baldus CR, Bridwell KH, Lenke LG, Okubadejo GO. Can we safely reduce blood loss during lumbar pedicle subtraction osteotomy procedures using tranexamic acid or aprotinin? A comparative study with controls. Spine (Phila Pa 1976). 2010 Jan 15;35(2):235-9. doi: 10.1097/BRS.0b013e3181c86cb9. PMID 20081519
- [Background] Daubs MD, Lenke LG, Cheh G, Stobbs G, Bridwell KH. Adult spinal deformity surgery: complications and outcomes in patients over age 60. Spine (Phila Pa 1976). 2007 Sep 15;32(20):2238-44. doi: 10.1097/BRS.0b013e31814cf24a. PMID 17873817
- [Background] Eck KR, Bridwell KH, Ungacta FF, Riew KD, Lapp MA, Lenke LG, Baldus C, Blanke K. Complications and results of long adult deformity fusions down to l4, l5, and the sacrum. Spine (Phila Pa 1976). 2001 May 1;26(9):E182-92. doi: 10.1097/00007632-200105010-00012. PMID 11337635
- [Background] La Maida GA, Luceri F, Gallozzi F, Ferraro M, Bernardo M. Complication rate in adult deformity surgical treatment: safety of the posterior osteotomies. Eur Spine J. 2015 Nov;24 Suppl 7:879-86. doi: 10.1007/s00586-015-4275-5. Epub 2015 Oct 6. PMID 26443695
- [Background] Lafage V, Smith JS, Bess S, Schwab FJ, Ames CP, Klineberg E, Arlet V, Hostin R, Burton DC, Shaffrey CI; International Spine Study Group. Sagittal spino-pelvic alignment failures following three column thoracic osteotomy for adult spinal deformity. Eur Spine J. 2012 Apr;21(4):698-704. doi: 10.1007/s00586-011-1967-3. Epub 2011 Aug 12. PMID 21837411
- [Background] Lee SH, Kim KT, Suk KS, Lee JH, Seo EM, Huh DS. Sagittal decompensation after corrective osteotomy for lumbar degenerative kyphosis: classification and risk factors. Spine (Phila Pa 1976). 2011 Apr 15;36(8):E538-44. doi: 10.1097/BRS.0b013e3181f45a17. PMID 21240054
- [Background] Iki M. [Epidemiology of osteoporosis in Japan]. Clin Calcium. 2012 Jun;22(6):797-803. Japanese. PMID 22653016
- [Background] Orimo H, Hashimoto T, Sakata K, Yoshimura N, Suzuki T, Hosoi T. Trends in the incidence of hip fracture in Japan, 1987-1997: the third nationwide survey. J Bone Miner Metab. 2000;18(3):126-31. doi: 10.1007/pl00010636. PMID 10783845
- [Background] Fujibayashi S, Hynes RA, Otsuki B, Kimura H, Takemoto M, Matsuda S. Effect of indirect neural decompression through oblique lateral interbody fusion for degenerative lumbar disease. Spine (Phila Pa 1976). 2015 Feb 1;40(3):E175-82. doi: 10.1097/BRS.0000000000000703. PMID 25394317
- [Background] Bridwell KH, Lewis SJ, Lenke LG, Baldus C, Blanke K. Pedicle subtraction osteotomy for the treatment of fixed sagittal imbalance. J Bone Joint Surg Am. 2003 Mar;85(3):454-63. doi: 10.2106/00004623-200303000-00009. PMID 12637431
- [Background] Cho SK, Bridwell KH, Lenke LG, Cho W, Zebala LP, Pahys JM, Kang MM, Yi JS, Baldus CR. Comparative analysis of clinical outcome and complications in primary versus revision adult scoliosis surgery. Spine (Phila Pa 1976). 2012 Mar 1;37(5):393-401. doi: 10.1097/BRS.0b013e31821f0126. PMID 21540777
- [Background] Dorward IG, Lenke LG, Bridwell KH, O'Leary PT, Stoker GE, Pahys JM, Kang MM, Sides BA, Koester LA. Transforaminal versus anterior lumbar interbody fusion in long deformity constructs: a matched cohort analysis. Spine (Phila Pa 1976). 2013 May 20;38(12):E755-62. doi: 10.1097/BRS.0b013e31828d6ca3. PMID 23442780
- [Background] Salvi G, Aubin CE, Le Naveaux F, Wang X, Parent S. Biomechanical analysis of Ponte and pedicle subtraction osteotomies for the surgical correction of kyphotic deformities. Eur Spine J. 2016 Aug;25(8):2452-60. doi: 10.1007/s00586-015-4279-1. Epub 2015 Oct 14. PMID 26467339
- [Background] Berjano P, Cecchinato R, Sinigaglia A, Damilano M, Ismael MF, Martini C, Villafane JH, Lamartina C. Anterior column realignment from a lateral approach for the treatment of severe sagittal imbalance: a retrospective radiographic study. Eur Spine J. 2015 Apr;24 Suppl 3:433-8. doi: 10.1007/s00586-015-3930-1. Epub 2015 Apr 17. PMID 25893333
- [Background] Bridwell KH, Lewis SJ, Edwards C, Lenke LG, Iffrig TM, Berra A, Baldus C, Blanke K. Complications and outcomes of pedicle subtraction osteotomies for fixed sagittal imbalance. Spine (Phila Pa 1976). 2003 Sep 15;28(18):2093-101. doi: 10.1097/01.BRS.0000090891.60232.70. PMID 14501920
- [Background] Kim YJ, Bridwell KH, Lenke LG, Rhim S, Cheh G. Pseudarthrosis in long adult spinal deformity instrumentation and fusion to the sacrum: prevalence and risk factor analysis of 144 cases. Spine (Phila Pa 1976). 2006 Sep 15;31(20):2329-36. doi: 10.1097/01.brs.0000238968.82799.d9. PMID 16985461
- [Background] Kim YJ, Bridwell KH, Lenke LG, Rinella AS, Edwards C 2nd. Pseudarthrosis in primary fusions for adult idiopathic scoliosis: incidence, risk factors, and outcome analysis. Spine (Phila Pa 1976). 2005 Feb 15;30(4):468-74. doi: 10.1097/01.brs.0000153392.74639.ea. PMID 15706346
- [Background] Annis P, Lawrence BD, Spiker WR, Zhang Y, Chen W, Daubs MD, Brodke DS. Predictive factors for acute proximal junctional failure after adult deformity surgery with upper instrumented vertebrae in the thoracolumbar spine. Evid Based Spine Care J. 2014 Oct;5(2):160-2. doi: 10.1055/s-0034-1386755. PMID 25278891
- [Background] Daubs MD. Sagittal alignment changes and proximal junctional kyphosis in adolescent idiopathic scoliosis. Spine J. 2016 Jun;16(6):784-5. doi: 10.1016/j.spinee.2016.02.019. PMID 27342708
- [Background] Fujimori T, Inoue S, Le H, Schairer WW, Berven SH, Tay BK, Deviren V, Burch S, Iwasaki M, Hu SS. Long fusion from sacrum to thoracic spine for adult spinal deformity with sagittal imbalance: upper versus lower thoracic spine as site of upper instrumented vertebra. Neurosurg Focus. 2014 May;36(5):E9. doi: 10.3171/2014.3.FOCUS13541. PMID 24785491
- [Background] Glassman SD, Coseo MP, Carreon LY. Sagittal balance is more than just alignment: why PJK remains an unresolved problem. Scoliosis Spinal Disord. 2016 Jan 22;11:1. doi: 10.1186/s13013-016-0064-0. eCollection 2016. PMID 27252982
- [Background] Glattes RC, Bridwell KH, Lenke LG, Kim YJ, Rinella A, Edwards C 2nd. Proximal junctional kyphosis in adult spinal deformity following long instrumented posterior spinal fusion: incidence, outcomes, and risk factor analysis. Spine (Phila Pa 1976). 2005 Jul 15;30(14):1643-9. doi: 10.1097/01.brs.0000169451.76359.49. PMID 16025035
- [Background] Hyun SJ, Kim YJ, Rhim SC. Patients with proximal junctional kyphosis after stopping at thoracolumbar junction have lower muscularity, fatty degeneration at the thoracolumbar area. Spine J. 2016 Sep;16(9):1095-101. doi: 10.1016/j.spinee.2016.05.008. Epub 2016 May 20. PMID 27217332
- [Background] Inoue S, Khashan M, Fujimori T, Berven SH. Analysis of mechanical failure associated with reoperation in spinal fusion to the sacrum in adult spinal deformity. J Orthop Sci. 2015 Jul;20(4):609-16. doi: 10.1007/s00776-015-0729-1. Epub 2015 May 12. PMID 25963608
- [Background] Kim HJ, Bridwell KH, Lenke LG, Park MS, Song KS, Piyaskulkaew C, Chuntarapas T. Patients with proximal junctional kyphosis requiring revision surgery have higher postoperative lumbar lordosis and larger sagittal balance corrections. Spine (Phila Pa 1976). 2014 Apr 20;39(9):E576-80. doi: 10.1097/BRS.0000000000000246. PMID 24480958
- [Background] Kim HJ, Yagi M, Nyugen J, Cunningham ME, Boachie-Adjei O. Combined anterior-posterior surgery is the most important risk factor for developing proximal junctional kyphosis in idiopathic scoliosis. Clin Orthop Relat Res. 2012 Jun;470(6):1633-9. doi: 10.1007/s11999-011-2179-1. PMID 22086507
- [Background] Kim YC, Lenke LG, Bridwell KH, Hyun SJ, You KH, Kim YW, Chang HG, Kelly MP, Koester LA, Blanke KM, Bumpass DB. Results of Revision Surgery for Proximal Junctional Kyphosis Following Posterior Segmental Instrumentation: Minimum 2-Year Postrevision Follow-Up. Spine (Phila Pa 1976). 2016 Dec 15;41(24):E1444-E1452. doi: 10.1097/BRS.0000000000001664. PMID 27128389
- [Background] Kim YJ, Bridwell KH, Lenke LG, Kim J, Cho SK. Proximal junctional kyphosis in adolescent idiopathic scoliosis following segmental posterior spinal instrumentation and fusion: minimum 5-year follow-up. Spine (Phila Pa 1976). 2005 Sep 15;30(18):2045-50. doi: 10.1097/01.brs.0000179084.45839.ad. PMID 16166893
- [Background] Lau D, Funao H, Clark AJ, Nicholls F, Smith J, Bess S, Shaffrey C, Schwab FJ, Lafage V, Deviren V, Hart R, Kebaish KM, Ames CP; International Spine Study Group. The Clinical Correlation of the Hart-ISSG Proximal Junctional Kyphosis Severity Scale With Health-Related Quality-of-life Outcomes and Need for Revision Surgery. Spine (Phila Pa 1976). 2016 Feb;41(3):213-23. doi: 10.1097/BRS.0000000000001326. PMID 26641842
- [Background] Park SJ, Lee CS, Chung SS, Lee JY, Kang SS, Park SH. Different Risk Factors of Proximal Junctional Kyphosis and Proximal Junctional Failure Following Long Instrumented Fusion to the Sacrum for Adult Spinal Deformity: Survivorship Analysis of 160 Patients. Neurosurgery. 2017 Feb 1;80(2):279-286. doi: 10.1227/NEU.0000000000001240. PMID 28173513
- [Background] Scheer JK, Osorio JA, Smith JS, Schwab F, Lafage V, Hart RA, Bess S, Line B, Diebo BG, Protopsaltis TS, Jain A, Ailon T, Burton DC, Shaffrey CI, Klineberg E, Ames CP; International Spine Study Group. Development of Validated Computer-based Preoperative Predictive Model for Proximal Junction Failure (PJF) or Clinically Significant PJK With 86% Accuracy Based on 510 ASD Patients With 2-year Follow-up. Spine (Phila Pa 1976). 2016 Nov 15;41(22):E1328-E1335. doi: 10.1097/BRS.0000000000001598. PMID 27831987
- [Background] Wang H, Ma L, Yang D, Wang T, Yang S, Wang Y, Wang Q, Zhang F, Ding W. Incidence and risk factors for the progression of proximal junctional kyphosis in degenerative lumbar scoliosis following long instrumented posterior spinal fusion. Medicine (Baltimore). 2016 Aug;95(32):e4443. doi: 10.1097/MD.0000000000004443. PMID 27512860
- [Background] Wu JC, Tang CT, Wu DL, Tsai TH, Chiang YH. Treatment of adjacent vertebral fractures following multiple-level spinal fusion. Acta Neurochir Suppl. 2008;101:153-5. doi: 10.1007/978-3-211-78205-7_26. PMID 18642651
- [Background] Yan P, Bao H, Qiu Y, Bao M, Varghese JJ, Sun X, Liu Z, Zhu Z, Qian B, Zheng M, Zhu F. Mismatch Between Proximal Rod Contouring and Proximal Junctional Angle: A Predisposed Risk Factor for Proximal Junctional Kyphosis in Degenerative Scoliosis. Spine (Phila Pa 1976). 2017 Mar;42(5):E280-E287. doi: 10.1097/BRS.0000000000001883. PMID 27557450
- [Background] Lenke LG, Fehlings MG, Shaffrey CI, Cheung KM, Carreon L, Dekutoski MB, Schwab FJ, Boachie-Adjei O, Kebaish KM, Ames CP, Qiu Y, Matsuyama Y, Dahl BT, Mehdian H, Pellise-Urquiza F, Lewis SJ, Berven SH. Neurologic Outcomes of Complex Adult Spinal Deformity Surgery: Results of the Prospective, Multicenter Scoli-RISK-1 Study. Spine (Phila Pa 1976). 2016 Feb;41(3):204-12. doi: 10.1097/BRS.0000000000001338. PMID 26866736
- [Background] Buchowski JM, Bridwell KH, Lenke LG, Kuhns CA, Lehman RA Jr, Kim YJ, Stewart D, Baldus C. Neurologic complications of lumbar pedicle subtraction osteotomy: a 10-year assessment. Spine (Phila Pa 1976). 2007 Sep 15;32(20):2245-52. doi: 10.1097/BRS.0b013e31814b2d52. PMID 17873818
- [Background] Fleischer GD, Kim YJ, Ferrara LA, Freeman AL, Boachie-Adjei O. Biomechanical analysis of sacral screw strain and range of motion in long posterior spinal fixation constructs: effects of lumbosacral fixation strategies in reducing sacral screw strains. Spine (Phila Pa 1976). 2012 Feb 1;37(3):E163-9. doi: 10.1097/BRS.0b013e31822ce9a7. PMID 21857409
- [Background] Tsuchiya K, Bridwell KH, Kuklo TR, Lenke LG, Baldus C. Minimum 5-year analysis of L5-S1 fusion using sacropelvic fixation (bilateral S1 and iliac screws) for spinal deformity. Spine (Phila Pa 1976). 2006 Feb 1;31(3):303-8. doi: 10.1097/01.brs.0000197193.81296.f1. PMID 16449903
- [Background] Bridwell KH, Edwards CC 2nd, Lenke LG. The pros and cons to saving the L5-S1 motion segment in a long scoliosis fusion construct. Spine (Phila Pa 1976). 2003 Oct 15;28(20):S234-42. doi: 10.1097/01.BRS.0000092462.45111.27. PMID 14560197
- [Background] Edwards CC 2nd, Bridwell KH, Patel A, Rinella AS, Berra A, Lenke LG. Long adult deformity fusions to L5 and the sacrum. A matched cohort analysis. Spine (Phila Pa 1976). 2004 Sep 15;29(18):1996-2005. doi: 10.1097/01.brs.0000138272.54896.33. PMID 15371700
- [Background] Gehrchen M, Hallager DW, Dahl B, Harris J, Gudipally M, Jenkins S, Wu AM, Bucklen BS. Rod Strain After Pedicle Subtraction Osteotomy: A Biomechanical Study. Spine (Phila Pa 1976). 2016 Apr;41 Suppl 7:S24. doi: 10.1097/BRS.0000000000001431. PMID 27015065
- [Background] Kim YJ, Bridwell KH, Lenke LG, Rhim S, Kim YW. Is the T9, T11, or L1 the more reliable proximal level after adult lumbar or lumbosacral instrumented fusion to L5 or S1? Spine (Phila Pa 1976). 2007 Nov 15;32(24):2653-61. doi: 10.1097/BRS.0b013e31815a5a9d. PMID 18007240
- [Background] Kuhns CA, Bridwell KH, Lenke LG, Amor C, Lehman RA, Buchowski JM, Edwards C 2nd, Christine B. Thoracolumbar deformity arthrodesis stopping at L5: fate of the L5-S1 disc, minimum 5-year follow-up. Spine (Phila Pa 1976). 2007 Nov 15;32(24):2771-6. doi: 10.1097/BRS.0b013e31815a7ece. PMID 18007259

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-12-04): https://cdn.clinicaltrials.gov/large-docs/09/NCT04536909/Prot_SAP_002.pdf
  • Informed Consent Form (2020-05-07): https://cdn.clinicaltrials.gov/large-docs/09/NCT04536909/ICF_001.pdf